CLINICAL TRIAL: NCT05285163
Title: The Effect of Palliative Care Training on Symptom Management, Rehospitalization and Quality of Life in Chronic Heart Failure: : A Randomized Controlled Trial
Brief Title: The Effect of Palliative Care Training on Symptom Management and Quality of Life in Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Gülşah Çamcı, Assistant Prof, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MU-SBF-IHH-GC-01
Record Dates: First submitted 2022-03-04; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure; End of Life
Keywords: heart failure; palliative care; rehospitalization; symptom burden; quality of life
MeSH Terms: conditions — Heart Failure; Death

STUDY DESIGN:
Intervention Model Description: The control group took usual care and the intervention group took both usual care and palliative care.
Who Masked: Participant
Masking Description: The patients were distributed with the minimization method of covariate-oriented randomization. According to NYHA (class III, IV), sex (male and female), and the number of hospitalizations (≤3 and ≥4) within one year, the patients were randomly appointed to the control and intervention groups. Thus, the patients in the intervention and control groups were distributed as homogeneous.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- palliative care education (Experimental): The patients in the intervention group were presented palliative care training in addition to their usual care. The training period lasts at least 45 minutes. After the training, patients were given the book 'Palliative Care in Heart Failure'. In this training, patients were informed about heart failure and pharmacological and non-pharmacological methods for symptoms such as dyspnea, pain, constipation, depression, edema, tiredness, nausea. The patients were followed up by telephone at the first, third, and sixth months after discharge. The patient's symptoms and quality of life were re-evaluated in telephone follow-up. During the follow-up period, the patient's training related to symptoms was repeated. The patients were referred to the physician for the symptoms and problems which they experienced in the house.
  Interventions: Behavioral: palliative care educatiom
- usual care (No Intervention): Firstly, the usual care provided to patients was described. It was determined that patients were not given regular and comprehensive training on heart failure, and no training was given on palliative care. Written educational material was not given to the patients. Patients were not followed up after discharge. Palliative care was not discussed with patients and their relatives. Also, they were not asked about their preferences. In usual care, Heart failure patients received medical treatment for their symptoms during hospitalization.

INTERVENTIONS:
Behavioral: palliative care educatiom — The patients in the intervention group were presented palliative care training in addition to their usual care
  Arms: palliative care education

SUMMARY:
Palliative care is of great importance because of poor quality of life and high mortality risk in advanced heart failure. This study was planned as a randomized controlled trial to determine the effect of palliative care training on symptom management, rehospitalization, and quality of life among patients with heart failure.

DETAILED DESCRIPTION:
Patients were informed about the research and written informed consent was obtained. Data were collected by face-to-face interviews within two days before discharge. Patient information form and scales were applied to Patients in the intervention and control groups. Patients in the intervention group were received education after filling the forms. The training was given one by one at the hospital. One or two relatives of patients were included in the training. The patient was comfortably seated, and the room door was closed, face to face interaction was conducted. The patient and his/her relatives were allowed to ask questions during the training. The patient in the intervention group received at least 45 minutes of data collection from a case because of detailed training. It took about 15 minutes to collect data from a patient in the control group. In some patients, the training program was divided to be clearer. The patients were traced by telephone at the first, third, and sixth months after discharge. The investigator's phone number was presented to the patients and they were told that they could call at any time. Continuous communication was ensured by giving the educator's phone number to the patients. The training was repeated by contacting the phone. The intervention group was retrained about symptoms they experienced during their telephone interview. The training was given to the experimental group as planned. No modifications/changes were made to the intervention during the study. Special notes were taken for each patient. The effect of the education given on the quality of life and symptom management was evaluated with questionnaires. The intervention was adhered to as planned.

ELIGIBILITY:
Inclusion Criteria:

* 18-year-old or over,
* Class III and IV heart failure patients according to New York Heart Association (NYHA) classification,
* Patients without any communication problem to prevent participation in the research [loss of hearing, visual impairment, lack of understanding/speaking in Turkish], can be contacted by telephone, are literate.
* The patients who were diagnosed with heart failure at least six months ago accepted to participate voluntarily were also included in the study.

Exclusion Criteria:

* Patients who wish to quit their study voluntarily during the study period and patients who died or worsened during the study period.

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-11-10 (Actual)

PRIMARY OUTCOMES:
Edmonton symptom assessment scale | six months
  ESAS consists of 10 symptoms as tiredness, pain, feeling of well-being, nausea, depression, anxiety, lack of appetite, drowsiness, shortness of breath, and others. Each symptom is scored between 0 and 10. While Zero points indicate no symptoms, 10 points are severe of symptoms.

SECONDARY OUTCOMES:
LVD-36-left ventricular dysfunction questionnaire | six months
  The questionnaire consists of 36 questions and the questions are answered as true or false. The correct answers are collected and indicated as the total percentage. The score is 0-100. High scores indicate poor quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah Çamcı, PhD, Principal Investigator — Marmara University
Locations (2):
- Turkey (Türkiye) (2):
  - Marmara U., Istanbul
  - Marmara University, Istanbul

IPD SHARING:
Plan to Share IPD: No
After the article is published, the results of the study will be shared.